CLINICAL TRIAL: NCT03819296
Title: Role of Microbiome in the Realm of Immune-Checkpoint Inhibitor Induced GI Complications In Cancer Population
Brief Title: Role of Gut Microbiome and Fecal Transplant on Medication-Induced GI Complications in Patients With Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2018-0383; NCI-2018-03437 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2018-0383 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2019-01-25; First posted 2019-01-28 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2025-09

CONDITIONS: Clinical Stage 0 Cutaneous Melanoma AJCC v8; Clinical Stage I Cutaneous Melanoma AJCC v8; Clinical Stage IA Cutaneous Melanoma AJCC v8; Clinical Stage IB Cutaneous Melanoma AJCC v8; Clinical Stage II Cutaneous Melanoma AJCC v8; Clinical Stage IIA Cutaneous Melanoma AJCC v8; Clinical Stage IIB Cutaneous Melanoma AJCC v8; Clinical Stage IIC Cutaneous Melanoma AJCC v8; Clinical Stage III Cutaneous Melanoma AJCC v8; Clinical Stage IV Cutaneous Melanoma AJCC v8; Colitis; Lung Non-Small Cell Carcinoma; Malignant Genitourinary System Neoplasm; Malignant Solid Neoplasm; Pathologic Stage 0 Cutaneous Melanoma AJCC v8; Pathologic Stage I Cutaneous Melanoma AJCC v8; Pathologic Stage IA Cutaneous Melanoma AJCC v8; Pathologic Stage IB Cutaneous Melanoma AJCC v8; Pathologic Stage II Cutaneous Melanoma AJCC v8; Pathologic Stage IIA Cutaneous Melanoma AJCC v8; Pathologic Stage IIB Cutaneous Melanoma AJCC v8; Pathologic Stage IIC Cutaneous Melanoma AJCC v8; Pathologic Stage III Cutaneous Melanoma AJCC v8; Pathologic Stage IIIA Cutaneous Melanoma AJCC v8; Pathologic Stage IIIB Cutaneous Melanoma AJCC v8; Pathologic Stage IIIC Cutaneous Melanoma AJCC v8; Pathologic Stage IIID Cutaneous Melanoma AJCC v8; Pathologic Stage IV Cutaneous Melanoma AJCC v8; Stage 0 Lung Cancer AJCC v8; Stage I Lung Cancer AJCC v8; Stage IA1 Lung Cancer AJCC v8; Stage IA2 Lung Cancer AJCC v8; Stage IA3 Lung Cancer AJCC v8; Stage IB Lung Cancer AJCC v8; Stage II Lung Cancer AJCC v8; Stage IIA Lung Cancer AJCC v8; Stage IIB Lung Cancer AJCC v8; Stage III Lung Cancer AJCC v8; Stage IIIA Lung Cancer AJCC v8; Stage IIIB Lung Cancer AJCC v8; Stage IIIC Lung Cancer AJCC v8; Stage IV Lung Cancer AJCC v8; Stage IVA Lung Cancer AJCC v8; Stage IVB Lung Cancer AJCC v8
MeSH Terms: conditions — Colitis; Carcinoma, Non-Small-Cell Lung; Urogenital Neoplasms; Lung Neoplasms | interventions — Practice Guidelines as Topic; Standard of Care; Endoscopy; Fecal Microbiota Transplantation; Infliximab; CT-P13; Prednisone; deltacortene; prednylidene; vedolizumab; Immunoglobulin G; Disulfides; LDP-02

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Supportive Care (standard of care, sample collection, FMT) (Experimental): PROJECT 1: Patients receive standard of care and undergo collection of stool and blood samples.
  PROJECT 2: Patients receive prednisone, infliximab, or vedolizumab per standard of care and undergo standard of care endoscopy 2 months after treatment. Patients also undergo collection of stool, blood, and tissue samples.
  PROJECT 3: Patients undergo FMT.
  Interventions: Other: Best Practice; Other: Biospecimen Collection; Procedure: Endoscopic Procedure; Procedure: Fecal Microbiota Transplantation; Biological: Infliximab; Other: Laboratory Biomarker Analysis; Drug: Prednisone; Biological: Vedolizumab

INTERVENTIONS:
Other: Best Practice — Receive standard of care
  Other Names: standard of care; standard therapy
Other: Biospecimen Collection — Undergo collection of stool, blood, and tissue samples
Procedure: Endoscopic Procedure — Undergo endoscopy
  Other Names: Endoscopic Examination; Endoscopy
Procedure: Fecal Microbiota Transplantation — Undergo FMT
  Other Names: Fecal Material Transplantation; Fecal Transplantation; FMT; Poo Transplant; Poop Transplant; Stool Transplant
Biological: Infliximab — Given intravenously (IV)
  Other Names: Avakine; cA2; Remicade; Remsima
Other: Laboratory Biomarker Analysis — Ancillary studies
Drug: Prednisone — Given orally
  Other Names: .delta.1-Cortisone; 1, 2-Dehydrocortisone; Adasone; Cortancyl; Dacortin; DeCortin; Decortisyl; Decorton; Delta 1-Cortisone; Delta-Dome; Deltacortene; Deltacortisone; Deltadehydrocortisone; Deltasone; Deltison; Deltra; Econosone; Lisacort; Meprosona-F; Metacortandracin; Meticorten; Ofisolona; Orasone; Panafcort; Panasol-S; Paracort; Perrigo Prednisone; PRED; Predicor; Predicorten; Prednicen-M; Prednicort; Prednidib; Prednilonga; Predniment; Prednisone Intensol; Prednisonum; Prednitone; Promifen; Rayos; Servisone; SK-Prednisone
Biological: Vedolizumab — Given IV
  Other Names: Entyvio; Immunoglobulin G1, anti-(human integrin LPAM-1 (lymphocyte Peyer''s patch adhesion molecule 1)) (human-Mus musculus heavy chain), disulfide with human-Mus musculus kappa-chain, dimer; LDP 02; LDP-02; LDP02; MLN0002; MLN02

SUMMARY:
This trial studies the role of the gut microbiome and effectiveness of a fecal transplant on medication-induced gastrointestinal (GI) complications in patients with melanoma or genitourinary cancer. The gut microbiome (the bacteria and microorganisms that live in the digestive system) may affect whether or not someone develops colitis (inflammation of the intestines) during cancer treatment with immune-checkpoint inhibitor drugs. Studying samples of stool, blood, and tissue from patients with melanoma or genitourinary cancer may help doctors learn more about the effects of treatment on cells, and help doctors understand how well patients respond to treatment. Treatment with fecal transplantation may help to improve diarrhea and colitis symptoms.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To compare the difference in stool microbiome pattern between patients who develop immune-checkpoint inhibitor (ICPI)-related colitis and patients who don't develop ICPI-related colitis.

II. To compare the difference in stool microbiome pattern in patients who developed ICPI-related colitis before and after colitis medical treatment.

III. To assess the safety and tolerability and efficacy of fecal microbiota transplantation (FMT).

SECONDARY OBJECTIVES:

I. To identify and characterize immune profile and genetic factors associated with onset of ICPI-related colitis in blood and colon tissue.

II. To identify and characterize immune profile and genetic factors in blood and colon tissue that are associated with quick response of ICPI-related colitis to medical treatment.

III. To characterize the endoscopic and histologic features of ICPI-related colitis before and after medical treatment.

IV. To document the changes of ICPI-related symptoms and the impact on functioning and quality of life (QoL) from fecal microbiota transplantation by patient-reported outcomes (PRO).

V. To assess stool microbiome and cytokine features that are associated with good response to fecal microbiota transplantation.

VI. To assess the factors in genetic/immune profile obtained from blood and colon tissue that are associated with good response to fecal microbiota transplantation.

VII. To characterize the endoscopic and histologic features of ICPI-related colitis before and after fecal microbiota transplantation.

EXPLORATORY OBJECTIVES:

I. To identify and characterize immune profile and genetic factors associated with onset of ICPI-related colitis in inflamed colonic mucosa and its matched normal mucosa.

II. To characterize the immune profile and genetic factors from the colon tissue in these colitis patients among different histological subtypes.

III. To assess the pattern of stool microbiome that is associated with good tumor response to ICPI treatment.

IV. To assess the association between stool inflammatory markers (i.e. lactoferrin and calprotectin) and the severity of endoscopic/histologic inflammation.

V. To assess the sensitivity and specificity of stool inflammatory markers (i.e. lactoferrin and calprotectin) as an indicators of ICPI-relate colitis response to treatment.

VI. To assess the microbiome pattern that triggers the infections on immunosuppressant treatment for ICPI colitis.

OUTLINE:

PROJECT 1: Patients receive standard of care and undergo collection of stool and blood samples.

PROJECT 2: Patients receive prednisone, infliximab, or vedolizumab per standard of care and undergo standard of care endoscopy 2 months after treatment. Patients also undergo collection of stool, blood, and tissue samples.

PROJECT 3: Patients undergo fecal microbiota transplant (FMT).

After completion of study, patients are followed up periodically.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of any stage melanoma, Non-Small Cell Lung Cancer or genitourinary (GU) malignancies (Project 1).
2. Diagnosis of any cancer type (Projects 2 and 3)
3. Treatment with any ICPI agent
4. Ability to understand and willingness to sign an informed consent form and rate surveys
5. Life expectancy > 4 months (Project 3)
6. ICPI-related diarrhea and/or colitis of any grade with or without concurrent non- GI toxicity as the toxicity group (project 1)
7. Patients with no organ toxicity as the control group (project 1)
8. ICPI-related colitis and/or diarrhea of grade ≥ 2 as GI toxicity (initial episode or recurrence) receiving standard treatment of immunosuppressive agents (steroid, infliximab, vedolizumab, or ustekinumab) any time during the colitis disease course until sustained resolution of GI toxicity, or one- year time point after enrollment (Project 2)
9. ICPI-related colitis and/or diarrhea of grade ≥ 2 as GI toxicity without involvement of non- GI toxicity within 45 days prior to FMT (Project 3)
10. ICPI-related colitis and/or diarrhea of grade ≥ 2 within 45 days prior to FMT with ANY of the following characteristics (project 3):

    (i) refractory to treatment of steroid and two doses of non-steroidal immunosuppressants e.g. infliximab, vedolizumab or ustekinumab,

    (ii) contraindication for immunosuppressive treatment,

    (iii) recurrence after successful initial treatment,

    (iv) recurrent symptoms once steroid is tapered down/off or diarrhea/colitis symptoms are steroid dependent, or

    (v) patients with a history of refractory ICPI-related colitis and/or diarrhea to medical treatment, even if they have improved symptoms from supportive care within 45 days prior to FMT
11. No concern for active concomitant GI infection for the ICPI diarrhea/colitis work up at the time of protocol therapy initiation as confirmed by stool tests or as per the treating physician based on clinical presentation (project 3)
12. Patient who has been cleared for enrollment by Infectious Diseases consultant or treating physician if positive infection workup or screening tests (e.g. lifelong positive T-spot due to BCG inoculation, chronic colonization) prior to initiation of diarrhea/colitis treatment (project 3)

Exclusion Criteria:

1. Age younger than 18 years
2. History of inflammatory bowel disease, and/or radiation enteritis or colitis with active disease status at the time of study treatment initiation
3. Pregnant and breastfeeding women
4. Women of child-bearing potential who have positive urine or serum pregnancy test or refuse to do pregnancy test unless last menstrual cycle was > 1 year prior to consent and/ or clear documentation states that patient is peri- or post-menopausal or there was recent supporting objective evidence of 'no pregnancy' status (e.g. blood or imaging) within 30 days prior to date of study treatment
5. Patients who develop concurrent non- GI toxicity at the time of FMT treatment (project 3)
6. Patients with active bacterial or fungal infection (Project 3)
7. Donors at risk for monkeypox infection and/ or exposure as determined by a questionnaire (Project 3)

Withdrawal Criteria

1. Patients may withdraw from the trial at any time
2. Patients who develop GI perforation or toxic colitis that require surgery from ICPI colitis
3. In project 3, if the first 30% of cases fail the fecal transplant treatment, then project 3 will be terminated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2021-02-21 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Difference in stool microbiome pattern | Up to 1 year
  The primary endpoint is alpha diversity of bacteria species (measured using inverse Simpson index). It is a measure of diversity which takes into account the number of species present, as well as the relative abundance of each species. As species richness and evenness increase, so diversity increases.
Incidence of adverse events (AE) of fecal microbiota transplantation (FMT) (Project 3) | Up to 1 year
  Adverse events will be recorded by Common Terminology Criteria for Adverse Events version 5 as well as FMT-specific events. All events will be recorded with grade and attribution to FMT. Adverse events that are related to fecal microbiota transplantation will be summarized using frequency and percentage by AE grade, type and attributions.

SECONDARY OUTCOMES:
Immune profile factors associated with onset of ICPI-related colitis in blood and colon tissue | Up to 1 year
  Immunohistochemistry study for inflammatory markers will be performed on colon biopsies to measure the change in pattern after treatment. Blood and stool samples will be compared before and after immunosuppressive treatment longitudinally and also horizontally between quick response patients and slow/refractory patient.
Genetic factors associated with onset of ICPI-related colitis in blood and colon tissue | Up to 1 year
  Genomic bacterial DNA will be extracted from fecal samples, with the addition of a bead-beating lysis step. Genomic 16S ribosomal-RNA V4 variable region will be amplified and sequenced on the Illumina MiSeq platform to obtain the microbiome structure and composition.
Endoscopic and histologic features of ICPI-related colitis before and after medical treatment | Baseline up to 1 year
  We will assess the resolution of the following endoscopic presentations of ICPI-related colitis including large, deep ulcerations, erosions, diffuse or patchy erythema, inflammatory exudate, loss of vascular pattern, aphthae, and edema after medical treatment.
  We will assess the resolution of the following histological features of acute colitis and lymphocytic colitis including neutrophilic infiltration, cryptitis, crypt abscess, eosinophilia, intraepithelial apoptosis, and increased intraepithelial lymphocytic infiltration after medical treatment.
Changes of ICPI-related symptoms | Up to 1 year
  We will use MD Anderson Symptom Inventory (MDASI)-Colitis module to capture ICPI-related symptoms, which include 22 physical, psychological, and cognitive symptoms and colitis related symptoms. The ratings are on 0-10 numeric scales, ranging from "not present" to "as bad as you can imagine.
Changes of quality of life (QoL) | Up to 1 year
  MD Anderson Symptom Inventory (MDASI)-Colitis module includes 6 symptom interference items which could capture the impact of therapy on patient's physical and affective functioning. The ratings are on 0-10 numeric scales, ranging from "did not interfere " to "interfered completely ".
Cytokine features that are associated with good response to FMT | Up to 1 year
  We will compare the levels of many cytokines/chemokines by Luminex assays including IL-6, IL-17A, TNF-α, etc. between patients with good response and poor response to FMT.
Genetic factors associated with onset of ICPI-related colitis in blood and colon tissue | Up to 1 year
  Genomic bacterial DNA will be extracted from fecal samples, with the addition of a bead-beating lysis step. Genomic 16S ribosomal-RNA V4 variable region will be amplified and sequenced on the Illumina MiSeq platform to obtain the microbiome structure and composition. We will evaluate these factors between patients with good response and poor response to FMT.
Changes of endoscopic and histologic features of ICPI-related colitis before and after fecal microbiota transplantation | Baseline up to 1 year
  We will assess the resolution of the following endoscopic presentations of ICPI-related colitis including large, deep ulcerations, erosions, diffuse or patchy erythema, inflammatory exudate, loss of vascular pattern, aphthae, and edema after FMT.
  We will assess the resolution of the following histological features of acute colitis and lymphocytic colitis including neutrophilic infiltration, cryptitis, crypt abscess, eosinophilia, intraepithelial apoptosis, and increased intraepithelial lymphocytic infiltration after FMT.

CONTACTS AND LOCATIONS:
Overall Officials: Yinghong Wang, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org